CLINICAL TRIAL: NCT00192686
Title: Cultures From Total Knee Arthroplasties, Obtained a.m. Kamme-Lindberg in Revision Cases.
Brief Title: Cultures a.m.Kamme-Lindbergh in Suspicion of Infected TKA
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-04-011-CP
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Total Knee Arthritis; Viral; Infection, Slow Virus
MeSH Terms: conditions — Infections

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Procedure: culture a.m. Kamme-Lindberg

SUMMARY:
Cultures from total knee arthroplasties, obtained a.m. Kamme-Lindberg in revision cases.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pedersen, MD, Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital, Denmark
Locations (1):
- Northern Orthopaedic Division, Clinic Farsoe, Aalborg University Hospital, Farsø, Northern Jutland, Denmark

REFERENCES:
- See also: Paper published on the findings from this study — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Citation&list_uids=16856967